CLINICAL TRIAL: NCT04516317
Title: Very Severe Malaria Treated by Intravenous Artesunate: Epidemiology, Management, Outcome and Prognostic
Brief Title: Very Severe Malaria Treated by Intravenous Artesunate
Acronym: Palustar
Status: Completed | Type: Observational
Sponsor: Dr Fabrice BRUNEEL (Other)
Responsible Party: Sponsor-Investigator, Dr Fabrice BRUNEEL, Investigator MD, Versailles Hospital
Organization: Versailles Hospital (Other)
Other Study IDs: P20/18_Palustar
Record Dates: First submitted 2020-07-09; First posted 2020-08-18 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Severe Malaria
Keywords: Severe Malaria; Artesunate; Critical Care; Quinine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group intravenous artesunate (around 300 patients): Period 2011-2019
  Interventions: Other: None (Observational study Group intravenous artesunate)
- Group intravenous quinine (around 300 patients): Period 2000-2010
  Interventions: Other: None (Observational study Group intravenous quinine)

INTERVENTIONS:
Other: None (Observational study Group intravenous artesunate) — Retrospective descriptive study of Group intravenous artesunate
  Groups: Group intravenous artesunate (around 300 patients)
Other: None (Observational study Group intravenous quinine) — Retrospective descriptive study of Group intravenous quinine
  Groups: Group intravenous quinine (around 300 patients)

SUMMARY:
In endemic areas, Plasmodium falciparum malaria exacts a huge public health toll, causing close to half a million deaths each year. In non-endemic industrialized areas, imported malaria may develop. In France, around 5000 imported cases occured annually, including 10-15% of severe malaria.

The criteria for defining severe malaria in endemic areas are established by the World Health Organization (WHO), and have been adjusted for severe imported malaria. In France, in order to optimize management, severe imported malaria is separated into two groups: very severe malaria (VSM) and less severe malaria (LSM). Briefly VSM included coma and/or shock and/or respiratory failure and/or acidosis and/or hyperlactatemia and/or death during hospitalization.

In France, severe imported malaria is treated with intravenous artesunate. Little is known about the management of imported VSM in the ICU with intravenous artesunate.

In a French national multicentric retrospective frame, the main objective of the present study is to describe in detail: epidemiology, management, outcome and prognostic of very severe imported malaria treated with intravenous artesunate during the period 2011-2019. The second objective is to retrospectively compare two groups : VSM treated with intravenous artesunate in the ICU during 2011-2019 versus VSM treated with intravenous quinine in the ICU during 2000-2010.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* More than 18 year-old at the time of inclusion AND
* Hospitalization in the ICU AND
* For severe imported malaria (Plasmodium falciparum) AND
* Very Severe Malaria episode defined during the 72 first hours as :

  * Neurological failure: Glasgow Coma Scale score<11 or repeated convulsions and/or
  * Shock: Systolic Blood Pressure<80 mmHg despite adequate fluid loading or need for vasoactive drugs and/or
  * Respiratory distress: Mechanical Ventilation or Non Invasive Ventilation ; or if spontaneous breathing: arterial pO2<60 mmHg or pulse oxymetry<92% in room air ; or Respiratory Rate>32/min and/or
  * Acidosis: plasma bicarbonate <15 mmol/l, or pH<7,35 and/or
  * Hyperlactatemia > 5 mmol/l and/or
  * Death during hospitalization for VSM

Exclusion Criteria:

* Less than 18 year-old at the time of inclusion OR
* Opposition to participate in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Very severe malaria in adults / Antimalarial treatment (Artesunate period 2011-2019 ; Quinine period 2000-2010)
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Mortality rate in the Group intravenous artesunate | At hospital discharge, an average of 1 month
  Mortality reported as a mortality rate (%)

SECONDARY OUTCOMES:
Mortality rates in the Group artesunate and Group quinine | At hospital discharge, an average of 1 month
  Mortality reported as a mortality rate (%)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice BRUNEEL, MD, Principal Investigator — Versailles Hospital Center
Locations (1):
- Fabrice BRUNEEL, Le Chesnay, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No